CLINICAL TRIAL: NCT02248077
Title: A Prospective, Randomized, Controlled, Multi-Center, Study Evaluating AutoloGel Therapy for Complete Closure of Wagner Grade 1-4 Diabetic Foot Ulcers, Venous Leg Ulcers and Stage II-IV Pressure Ulcers
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was redesigned in collaboration with CMS before it started.
Sponsor: Cytomedix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM-567
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Impaired Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AutoloGel (Active Comparator): AutoloGel consists of platelet-rich plasma (PRP) gel produced from the patient's own peripheral blood and pharmaceutical additives including calcium chloride, thrombin and ascorbic acid. The AutoloGel product is obtained by processing the patient's own blood using the AutoloGel System. After the final AutoloGel formulation is produced it is used immediately for patient's specific ulcer care.
  Interventions: Device: AutoloGel
- Usual and Customary Care (UCC) (Other): Standard of care
  Interventions: Other: Usual and Customary Care (UCC)

INTERVENTIONS:
Device: AutoloGel
  Arms: AutoloGel
Other: Usual and Customary Care (UCC)
  Arms: Usual and Customary Care (UCC)

SUMMARY:
This study is designed to demonstrate the outcome of complete ulcer closure of patients with Wagner Grade 1-4 DFUs, VLUs or Stage II-IV PUs using AutoloGel versus Usual and Customary Care (UCC).

ELIGIBILITY:
Inclusion Criteria:

For DFU indication:

1. Medicare beneficiary
2. Males or females ≥ 18 years of age
3. Type I or II diabetes requiring medical treatment as determined by the physician
4. The single wound to be applied Study Treatment (Index Ulcer) is a Wagner 1-4 DFU (see Section 17.12 Appendix 12 for Wagner Classification) that is located on the dorsal, plantar, medial, or lateral aspect of the foot (including all toe surfaces and the heel)
5. Patients have been treated with UCC at the center for 2 weeks prior to randomization with no greater than 20% reduction in wound area or volume and documented wound measurements are available
6. For patients with multiple potential Index DFUs, the largest ulcer will be selected. There must be at least 4 cm between the Index Ulcer and other ulcers; if all ulcers are closer than 4 cm, the patient should not be enrolled (screen failure)
7. Demonstrated offloading regimen
8. A wound age of ≥ 30 days at the Screening Visit
9. Patient must be willing to comply with the protocol, which will be assessed by enrolling clinician.
10. Patient must sign an Informed Consent Form prior to any study-related procedures.

For VLU indication:

1. Medicare beneficiary
2. Males or females ≥ 18 years of age
3. Diagnosed venous disease
4. Patients have been seen at the center/site for 2 weeks prior to randomization with no greater than 20% reduction in wound area or volume and documented wound measurements are available
5. The non-healing wound is located between the knee and ankle and may include ankle
6. For patients with multiple potential Index VLUs, the largest ulcer will be selected. There must be at least 4 cm between the Index Ulcer and other ulcers; if all ulcers are closer than 4 cm, the patient should not be enrolled (screen failure)
7. Demonstrated compression regimen
8. A wound age of ≥ 30 days at the Screening visit
9. Patient must be willing to comply with the protocol, which will be assessed by enrolling clinician
10. Patient must sign an Informed Consent prior to any study-related procedures.

For PU indication:

1. Medicare beneficiary
2. Males or females ≥ 18 years of age
3. Ulcer of pressure/shear etiology (Stage II, III, IV, see Section 17.13 Appendix 13 for stage definitions)
4. Patients have been seen at the site for 2 weeks prior to randomization with no greater than 20% reduction in wound area or volume and documented wound measurements are available
5. The single wound to be applied Study Treatment (Index Ulcer) that is located on the heel, ischium, sacrum, coccyx or trochanter
6. For patients with multiple potential PUs, the largest ulcer will be selected. There must be at least 4 cm between the Index Ulcer and other ulcers; if all ulcers are closer than 4 cm, the patient should not be enrolled (screen failure)
7. Demonstrated pressure relief regimen
8. A wound age of ≥ 30 days at Screening visit
9. Patient must be willing to comply with the Protocol, which will be assessed by enrolling clinician.
10. Patient must sign an Informed Consent prior to any study-related procedures.

Exclusion Criteria:

1. Patients known to be sensitive to AutoloGel components (calcium chloride, thrombin, ascorbic acid) and/or materials of bovine origin
2. Presence of another wound that is concurrently treated and might interfere with the treatment of the Index wound
3. Malignancy in wound bed
4. Active clinical wound infection.
5. Patient has inadequate venous access for repeated blood draw required for AutoloGel processing
6. Patients who are cognitively impaired and do not have a healthcare proxy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Complete Ulcer Closure | 12 weeks
  Proportion of patients with complete ulcer closure

REFERENCES:
- See also: Related Info — http://cytomedix.com